CLINICAL TRIAL: NCT01870128
Title: Comparison of Three Different Treatment Regimes in Early Rheumatoid Arthritis: A Randomized Open-labelled Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Atul Batra, Senio Resident, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T-54/ 12.06.2009
Record Dates: First submitted 2013-05-30; First posted 2013-06-05 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Steroid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methylprednisolone; Methotrexate; Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Methotrexate (Active Comparator): Single agent Methotrexate 15 to 25 mg PO per week
  Interventions: Drug: Methotrexate
- Combination (Active Comparator): Methotrexate 15 to 25 mg PO per week Hydroxychloroquine 200 mg Twice daily Sulfasalazine 2000 to 3000 mg per day
  Interventions: Drug: Combination
- Combination Steroid (Experimental): Methotrexate 15 to 25 mg PO per week Hydroxychloroquine 200 mg Twice daily Sulfasalazine 2000 to 3000 mg per day Methylprednisolone 1000 mg intravenous per day for 3 days
  Interventions: Drug: Combination Steroid

INTERVENTIONS:
Drug: Combination Steroid — Methylprednisolone 1000 mg intravenous for 3 days Methotrexate 15 to 25 mg PO per week Hydroxychloroquine 200 mg twice daily Sulfasalazine 2000 to 3000 mg per day
  Other Names: Methylprednisolone 1000 mg intravenous for 3 days
  Arms: Combination Steroid
Drug: Methotrexate — Methotrexate 15 to 25 mg PO per week
  Other Names: Methotrexate 15 to 25 mg PO per week
  Arms: Methotrexate
Drug: Combination — Methotrexate 15 to 25 mg PO per week Hydroxychloroquine 200 mg Twice daily Sulfasalazine 2000 to 3000 mg per day
  Other Names: Methotrexate 15 to 25 mg PO per week; Hydroxychloroquine 200 mg Twice daily; Sulfasalazine 2000 to 3000 mg per day
  Arms: Combination

SUMMARY:
Many studies have been conducted to evaluate the role of pulse steroids in early rheumatoid arthritis (RA) but no consensus exists. The aim of this study is to study the efficacy of various treatment regimens in early RA. Methods: This is a randomized open-labeled trial. Patients were randomised into three groups. In group A, patients were treated with single drug (methotrexate 15 mg/wk). The patients in Group B were treated with a combination of DMARDS (Methotrexate, sulfasalazine and hydroxychloroquine). The patients in Group C received combination therapy as in group B and 3 pulses of methylprednisolone intravenously.

DETAILED DESCRIPTION:
Many studies have been conducted to evaluate the role of pulse steroids in early rheumatoid arthritis (RA) but no consensus exists. The aim of this study is to study the efficacy of various treatment regimens in early RA. Patients were divided into three groups. In group A, patients were treated with single drug (methotrexate 15 mg/wk). The patients in Group B were treated with a combination of DMARDS (Methotrexate, sulfasalazine and hydroxychloroquine). The patients in Group C received combination therapy as in group B and 3 pulses of methylprednisolone intravenously.

ELIGIBILITY:
Inclusion Criteria:

1. Rheumatoid Arthritis diagnosed on the basis of revised American college of rheumatology criteria,1987
2. Age >18 years
3. Early Rheumatoid Arthritis i.e. less than 2 years duration
4. Patient giving consent to participate in study
5. Disease Modifying Anti-Rheumatic Drugs naive -

Exclusion Criteria:

1. Pregnant and lactating patient or planning to conceive in next year
2. Patient who had joint surgery in last 6 months
3. Co morbidities such as liver disease, kidney disease, hematological malignancies
4. Uncontrolled hypertension, diabetes mellitus
5. Coronary artery disease -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2009-08; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Response to treatment | 22 months
  To compare the response (EULAR criteria) to treatment in the three treatment groups.

SECONDARY OUTCOMES:
Disease activity score (DAS28) | 22 months
  To compare the disease activity score (DAS28) score and its defining variables (tender joint count, swollen joint count, erythrocyte sedimentation rate and patient global assessment on visual analogue scale).

CONTACTS AND LOCATIONS:
Overall Officials: ATUL BATRA, MD, Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- AIIMS, New Delhi, National Capital Territory of Delhi, India